CLINICAL TRIAL: NCT03835494
Title: Tissue Doppler Imaging - A Promising Technique To Assess Myocardial Function In Adult Fallot Patients
Brief Title: Analysis of RV-Dysfunction in Fallot Patients
Acronym: Fallot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Fallot
Record Dates: First submitted 2019-01-08; First posted 2019-02-08 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Tetralogy of Fallot
Keywords: Tetralogy of Fallot; Tissue Doppler Imaging; Exercise testing
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Intervention Model Description: Transthoracic echocardiography including TDI is performed at rest, during PLR, HG and CPX in Fallot patients and healthy controls. In Fallot patients, transthoracic ultrasound at rest and during CPX are part of the routinely follow-up. PLR and HG were performed additionally as part of the investigator's study to analyze TDI parameters during various endurance testings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fallot patients (Experimental): Fallot patients
  Interventions: Other: Transthoracic echocardiography at rest, during PLR, HG and CPX (including blood gas analysis in both groups). Additionally Fallot patients will undergo routine blood testings.
- healthy controls (Experimental): healthy volunteers
  Interventions: Other: Transthoracic echocardiography at rest, during PLR, HG and CPX (including blood gas analysis in both groups). Additionally Fallot patients will undergo routine blood testings.

INTERVENTIONS:
Other: Transthoracic echocardiography at rest, during PLR, HG and CPX (including blood gas analysis in both groups). Additionally Fallot patients will undergo routine blood testings. — Transthoracic echocardiography at rest, during PLR, HG and CPX (including blood gas analysis in both groups). Additionally Fallot patients will undergo routine blood testings.

SUMMARY:
In the presented study TDI will be used as a modern technique to characterize RV-function in Fallot patients at rest and during different exercise conditions.

DETAILED DESCRIPTION:
Tissue Doppler imaging (TDI) presents a modern technique to depict the velocity of tissue motion within a distinct area of the myocardium providing amendatory characterization of diastolic and systolic function of the heart. TDI is hypothesized to be of additional value in the evaluation of adult congenital heart disease, especially tetralogy of Fallot (TOF), which is one of the most common conditions. In particular, Fallot patients are at risk of developing right ventricular (RV) dysfunction due to pulmonary valve defects or alterations of the outflow tract. It is pivotal to recognize this progression at an early stage before irreversible changes occur. Aim of the study is to test feasibility of TDI in Fallot patients as a new technique that provides new parameters to characterize RV dysfunction, more precise than common methods. Additionally TDI is performed at rest and during different endurance testings (passive Leg Raising (PLR), handgrip (HG) and cardiopulmonary exercise (CPX), as certain changes might be compensated at rest, first apparent during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with corrected tetralogy of Fallot
* Adult healthy controls without cardiovascular disease or other relevant systemic diseases with written consent

Exclusion Criteria:

* Inability to give written consent, incapable of cycling or handgrip exercise due to cognitive or orthopedic limitation, poor echocardiographic image quality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Right ventricular myocardial velocity | Baseline
  Right ventricular myocardial velocity during early diastole (cm/s) Right ventricular myocardial velocity during late diastole (cm/s) Right ventricular myocardial velocity during systole (cm/s) baseline (one time point, measurements are performed at rest and during exercise)

SECONDARY OUTCOMES:
Peak oxygen consumption (ml/min/kg) and Oxygen consumption at anaerobic threshold (ml/min/kg) | Baseline
  CPX is performed for the measurement of TDI velocities at peak exercise, as well as for the assessment of the participants´ cardiopulmonary status. For the latter, the focus lies on oxygen consumption at peak exercise and at anaerobic threshold

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided